CLINICAL TRIAL: NCT06395935
Title: A Multi-center, Prospective, Randomized Study to Evaluate the Usefulness of Applying the Chronic Side Effect Management Platform (Wecare) in Gastric Cancer Survivors
Brief Title: Wecare Study in Gastric Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gyeongsang National University Hospital (Other)
Collaborators: National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Wecare2024
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional group (No Intervention): In the control group, participants will be asked to complete written questionnaires in the outpatient clinic before surgery and at 1, 3, and 6 months after surgery. Based on the questionnaires, a clinician will provide a solution at an outpatient clinic. However, the Wecare® platform was not provided. .
- Wecare group (Experimental): In the intervention group, participants will be asked to use the Wecare® platform (Figure 2). The Wecare® platform administers QoL questionnaires, including the KOQUSS-40 and EORTC QLQ-C30, following gastrectomy to treat gastric cancer. Based on participants' responses, The platform automatically generates expert recommendations from gastric cancer specialists based on participants' responses according to the timing of surgery after gastrectomy. Furthermore, the Wecare® platform offers educational materials on gastric cancer to address participants' questions about the disease. Participants will be free to use the platform but will be asked to visit the Wecare® platform at least once a month and answer questionnaires. Participants will visit an outpatient clinic before surgery and at 1, 3, and 6 months after surgery.
  Interventions: Other: Wecare (website)

INTERVENTIONS:
Other: Wecare (website) — support feedback of qutionaire & supply educational contents
  Arms: Wecare group

SUMMARY:
The KOrean QUality of life in Stomach cancer patients Study group (KOQUSS) made a method (KOQUSS-40) for assessing appropriately the quality of life of gastric cancer patients who have undergone gastrectomy, and developed a digital platform (Wecare) based on KOQUSS-40. In this study, we propose a randomized controlled trial to compare quality of life after gastrectomy in patients with and without smartphone app support.

DETAILED DESCRIPTION:
Smartphone apps have been gaining popularity in the delivery of lifestyle interventions in chronic disease management. In patients with cancer, randomized clinical trials have investigated the effect of smartphone-based interventions and reported improved quality of recovery and equal satisfaction with care compared with conventional in-person follow-up. However, there are no studies yet in which smartphone apps have evaluated the quality of life in patients after gastric cancer surgery.

Surgery is the mainstay of gastric cancer treatment. The proportion of patients with early gastric cancer and their survival rate of gastric cancer patients are increasing in East Asia thanks to the nationwide endoscopy screening program. As the number of long-term survivors after gastric cancer surgery increases, interest in the quality of life after surgery is also increasing. After gastrectomy, the remaining stomach volume is reduced or lost, and the vagus nerve is damaged during the surgery, which has various effects on the motor function and hormone secretion function of the stomach. Patients experience postgastrectomy syndrome, which includes lethargy, decreased appetite, early satiety, weight loss, abdominal distension, gastroesophageal reflux symptoms, diarrhea, anemia, and dumping syndrome. In addition to these physical symptoms, patients experience various symptoms and aftereffects after stomach cancer surgery, including psychological reactions such as fear, anxiety, and depression, and social problems such as avoidance of interpersonal relationships, social isolation, and difficulty returning to society.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (19-75 years) who underwent radical gastrectomy

Exclusion Criteria:

* Patients who were unable to undergo regular follow-up, lacked communication, or were deemed unsuitable to participate in this study by the researcher

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
the quality of life in gastric cancer survivor (KOQUSS-40) | at 1, 3, and 6 months after surgery in the outpatient clinic.
  KOQUSS-40 questionnaire has a 40-item questionnaire in 11 domains focusing on the symptoms evaluation after gastric cancer surgery.

SECONDARY OUTCOMES:
Weight | at 1, 3, and 6 months after surgery in the outpatient clinic.
  Weight change
nutritional index | at 1, 3, and 6 months after surgery in the outpatient clinic.
  nutritional index change
KOQUSS-40 questionnaire compliance | at 1, 3, and 6 months after surgery in the outpatient clinic.
  check the KOQUSS-40 questionnaire compliance

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Ho Jeong, MD, Principal Investigator — Gyeongsang National University Changwon Hospital
Locations (1):
- Gyeongsang National University Hospital, Changwon, Gyeongsandnam-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
if request, we can share the IPD without personal data.
Supporting Information: Study Protocol
Time Frame: The study was finished, the data can available
Access Criteria: Fore researcher, not for business model